CLINICAL TRIAL: NCT01682330
Title: The Long-term Effects of Training on Muscle Strength and Functionality
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s53571
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-06

CONDITIONS: Training; Ageing; Muscle Strength; Functionality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Fitness
- Whole-body vibration
- Control

SUMMARY:
The purpose of the present study is to evaluate the long-term effects of 1 year of high-intensity fitness training and low-intensity whole-body vibration training on muscle strength and functionality. Therefore, muscle strength and functionality are measured after a 6-yr interval in older adults (65+).

ELIGIBILITY:
Inclusion Criteria:

* female (+65 years)
* participation in previous study "De effecten van oefenprogramma's op gezondheids- en fitheidsgerelateerde parameters in een groep van 60-plussers" [The effects of exercise programs on health and fitness-related parameters in a group of people over 60]
* able to perform a maximal strength test on a dynamometer

Exclusion Criteria:

- pathologies that prohibit a maximal strength test on a dynamometer

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults (+65 years)
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)